CLINICAL TRIAL: NCT02339597
Title: Therapy Adherence in Different Settings of Automatic Positive Airway Pressure (APAP) Therapy Initiation in Patients With Obstructive Sleep Apnea (OSA): Comparison Between in Sleep-lab vs. at Home Environment.
Brief Title: Therapy Adherence of APAP Therapy Initiation in Sleep-lab Versus at Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Dr. Ingo Fietze (Other)
Collaborators: ResMed (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Ingo Fietze, Head of Sleep Lab, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EA1/306/13
Record Dates: First submitted 2014-01-27; First posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Patient Compliance
MeSH Terms: conditions — Patient Compliance | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- APAP Lab (Experimental): standard Initiation of APAP therapy in sleep laboratory.
  Interventions: Procedure: Automatic Positive Airway Pressure (APAP) initiation
- APAP Home (Experimental): initiation of APAP therapy in homely environment with additional continuous telemetric support.
  Interventions: Procedure: Automatic Positive Airway Pressure (APAP) initiation

INTERVENTIONS:
Procedure: Automatic Positive Airway Pressure (APAP) initiation

SUMMARY:
Primary hypothesis:

The objective compliance ( # of hours per night of APAP therapy) is higher in patients who get the APAP treatment initiation at home due to the fact that they get better support by telemetric control and the possibility of prompt interventions.

Secondary hypothesis:

Based on the higher support at the home APAP initiation the following parameters will be better in comparison to the standard supply in laboratory:

Objective measures:

* mask leakage
* pressure
* Apnea-Hypopnea-Index (AHI)

Subjective measures:

* quality of life
* sleepiness

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from patients after verbally and written informing
* Age between 18 and 80 Years
* obstructive sleep apnea syndrome (OSAS) with an AHI > 15/h and without previous therapy

Exclusion Criteria:

* Intolerance to wear the PAP therapy mask
* sleep breathing disorders (SBD) with central apneas > 20% and other sleep disorders
* disabilities who prevents the wear of a therapy mask
* initiated PAP therapy
* pre-treatment of OSAS incl. UPPP (uvulo palato pharyngo plasty)
* modified Mallampati Score T3 and T4
* participation on clinical studies 4 weeks before start of the study
* known or acute psychiatric/neurological or psychological disorders, who impairs the compliance to take part of the study.
* chronical or new clinically significant pneumological or cardiovascular disease (exception: effectively therapies of hypertension, cardiac arrhythmia and coronal cardiac disease)
* acute internistic disease
* neuromuscular disease
* condition after Apoplexy
* oncological disease in recent 5 years
* drug/alcohol consumption
* consumption of von psychotropic drugs, hypnotics and other drugs who are able to influence the sleep/wake cycle

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Number of usage hours of of positive airway pressure therapy per night | 6 month

SECONDARY OUTCOMES:
Apnea Hypopnea Index [1 / hour of sleep) | 6 month

OTHER OUTCOMES:
Quality of Life | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Charite-Universitaetsmedizin Berlin, Center for Sleep Medicine, Berlin, State of Berlin, Germany